CLINICAL TRIAL: NCT05587179
Title: The Impact of Different Recovery Positions on the Perfusion of the Lower Forearm and Comfort Associated With the Positioning: a Cross-over Randomized Controlled Trial
Brief Title: The Impact of Different Recovery Positions on the Perfusion of the Lower Forearm and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Evidence-Based Practice, Belgium (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RP-001
Record Dates: First submitted 2022-09-26; First posted 2022-10-19 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Unconsciousness
Keywords: Recovery position; First aid for unconsciousness; Arterial flow
MeSH Terms: conditions — Unconsciousness

STUDY DESIGN:
Intervention Model Description: This study is a cross-over Randomized Controlled Trial in which the sequence of the lateral recovery position will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral side-lying recovery position with extended arm (Experimental): The lateral side-lying recovery position with extended arm is directly based on the revised 2021 ERC guidelines recommending to extend the dependent arm and placing it next to the creased upper lying arm, which supports the head.
  Interventions: Other: recovery position
- Lateral side-lying recovery position with bent arms (Active Comparator): In the lateral side-lying recovery position with bent arms, the elbow of the dependent arm will now be bent with palm up and the far knee still flexed.
  Interventions: Other: recovery position

INTERVENTIONS:
Other: recovery position — A side-lying recovery position is a first aid intervention that can be performed by laypeople when victims are unresponsive but breathing normally and, hence, do not require cardiopulmonary resuscitation.

SUMMARY:
Introduction: A side-lying recovery position is recommended when victims are unresponsive but breathing normally and, hence, do not require cardiopulmonary resuscitation. In 2021, the European Resuscitation Council (ERC) and the Belgian Red Cross-Flanders issued new guidelines which included the description of a modified recovery position to avoid problems in victims with joint stiffness and to overcome potential obstructed venous return in the dependent arm. Based on good practice insights, the dependent arm will now be extended and not bent to support the other arm. However, there is currently no evidence available to support a specific recovery position.

Objectives: The aim of this study is to assess the impact of different recovery positions on perfusion of the forearm and associated comfort.

Methods: In this cross-over randomized controlled trial, 24 healthy volunteers will be placed in either the lateral recovery position with extended dependent arm or with bent arm, and in the other position thereafter. Before and between both recovery positions, the volunteers will be positioned supine for 15 min. Several perfusion indices of the forearm will be non-or mildly invasively monitored in the respective recovery positions by radial artery tonometry, ulnar artery echo doppler and venous congestion plethysmography. Subjective participant's discomfort and pain will be assessed as well. Differences in continuous outcomes between the different recovery positions will be assessed with paired t-tests or wilcoxon signed-rank test.

Discussion: The benefit of lateral positioning of adults and children with decreased level of consciousness has been widely accepted despite limited supportive scientific evidence. We here will provide direct evidence (i) whether venous drainage in the dependent limb is impaired when positioning the victim in the lateral recovery position with bent arms and (ii) whether this potential complication can be minimized by extending the dependent arm. The major limitations of this study is that healthy volunteers, instead of non-responsive victims, are included as participants, and that the study will be performed in a highly controlled environment. Nevertheless, the generated insights will directly fuel evidence-based treatment recommendations regarding the recovery position in first aid settings, and fill a current gap in evidence.

ELIGIBILITY:
Inclusion Criteria:

-healthy volunteers

Exclusion Criteria:

* History of any coronary or peripheral vascular disease such as Raynaud's disease or thromboangitis obliterans (self-declared)
* Type I or type II diabetes (self-declared)
* Intake of cholesterol-lowering medication (self-declared)
* High blood pressure (systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg) and/or use of antihypertensive drugs (self-declared)
* Obesity (BMI > 30 kg/m2)
* Smoking or using tobacco products (self-declared)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Difference in peripheral arterial pressure (PAP) | between 10 to 15 min in each position
  extracted from pulse wave amplitude (PWA) measured by radial artery tonometry
Cross-sectional area of the ulnar artery (SU) and peak systolic velocity of the ulnar artery (PSVU) of the hand of the dependent arm | between 10 to 15 min in each position
  measured by echo doppler
Peripheral venous pressure (PVP) | between 10 to 15 min in each position
  measured at the forearm and the back of the hand by venous congestion plethysmography

SECONDARY OUTCOMES:
Oxygen saturation | measured continuously during 1u15 min (15 min supine position, 15 min posture 1, 15 min supine position, 15 min posture 2, 15 min supine position)
Heart rate | measured continuously during 1u15min (15 min supine position, 15 min posture 1, 15 min supine position, 15 min posture 2, 15 min supine position)
Discomfort (experienced by participant) | after 15 min in the recovery position
  10-point Likert-scale completed by the participants
Pain (experienced by participant) | after 15 min in the recovery position
  10-point Likert-scale completed by the participants
Skin discoloration | after 15 min in the recovery position
  10-point Likert-scale completed by the researcher

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Heuten, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No